CLINICAL TRIAL: NCT06464471
Title: Comprehensive Health Assessment for My Plan: Implementation Study (CHAMP Implementation Study)
Brief Title: Comprehensive Health Assessment for My Plan: Initial Implementation Study (CHAMP Implementation Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other); Unity Health (Other)
Responsible Party: Principal Investigator, Martine Puts, Principal investigator, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CTO#4200
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Older Adults
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older adults completing the CHAMP tool before treatment decision is made (Experimental): Eligible participants who consent to the study will be asked to complete questionnaires about socio-demographic characteristics, literacy, and technology comfort. Subsequently, participants will be asked to complete the CHAMP tool at home or in the clinic before the participants' medical appointment with the clinician. Next, participants will see the clinician for the consultation. Approximately one week after the consultation, participants will be asked to complete 3 questionnaires about the participants' experience and satisfaction with the CHAMP tool.
  Interventions: Other: Self-reported online geriatric assessment (CHAMP)

INTERVENTIONS:
Other: Self-reported online geriatric assessment (CHAMP) — The CHAMP tool is a self reported online tool that has been developed to increase patients' accessibility to geriatric assessment and improve treatment decision making. The tool includes questions about function, mobility, cognition, nutrition, social support, depression substance use disorders, and miscellaneous items. Based on usability testing in the previous phase of this study, the tool can be completed in approximately 10-15 minutes. The tool generates a summary report with recommendations for patients and clinicians.

SUMMARY:
The current standard preoperative assessment does not consider the needs of older adults undergoing non-oncological surgery. To enhance the treatment decision-making and planning for older adult surgical patients, the British Geriatric Society and the American Society of Colon and Rectal Surgeons recommend the implementation of preoperative GA for all older adults. Geriatric assessment (GA) predicts treatment toxicity and overall mortality in older adults with complex health problems. However, in-person GA may not be feasible in several clinical settings for various reasons, including lack of training, time, or access to advanced geriatric services. These challenges can be minimized through a self-reported online GA that can be completed by patients prior to the participants' medical appointment. In a previous study, the investigators developed a self-reported online GA, known as the Comprehensive Health Assessment for My Cancer treatment Plan (CHAMP), which was used in geriatric oncology to increase accessibility to GA for older adults with cancer. In this study, the aim is to deploy the CHAMP tool to various clinics across 4 institutions and assess feasibility outcomes, as well as the efficacy of the CHAMP tool in the identification of geriatric issues and the development of supportive care.

DETAILED DESCRIPTION:
Introduction:

The aging population in Canada is greatly contributing to the growing number of older adults undergoing elective surgery. Approximately 48% of inpatient surgeries in Canada were aged at least 65 years old in 2021. Currently, the standard preoperative assessment does not include evaluations designed to address the needs of older adults. Increasing age is associated with changing physiology along with increasing comorbidity, polypharmacy, functional impairment, and cognitive impairment. Frailty (reduced physiologic reserve) is common but not universal. However, frailty in surgical settings vary between 13% to 84%, depending on the frailty evaluation tool used. Various systematic reviews have also identified an association between frailty and adverse events after surgery, including increased rates of postoperative complications, mortality, and discharge to a location other than home. The British Geriatric Society and the American Society of Colon and Rectal Surgeons thus recommend GA for OAs requiring non-oncological surgery. A GA has 8 key assessment domains (i.e. comorbidity, functional status, medications, falls risk, nutrition, social supports, cognition, mood), each of which is relevant to the "staging of the aging" and development of personalized treatment plans for older adults. In non-oncological surgery settings, GA can help reduce the risk of adverse outcomes of surgery, and optimize the health and functional status of older adults in the preoperative stage. However, GA has not been widely implemented in surgical settings due to the lack of time, training, and access to advanced geriatric services. An innovative, scalable solution is a patient self-completed electronic GA tool.

The investigators designed the CHAMP tool, a self-reported online GA that can be completed by older adults at home or in the clinic prior to the participants' medical appointment. The process for developing CHAMP included the following steps: i) a systematic review and a Delphi Panel of expert clinicians to select the final domains and items/questionnaires; ii) design sessions with older adults with cancer to develop the layout and contact of the tool; iii) usability sessions with older adults with cancer to finalize the tool; and iv) design sessions with oncology clinicians to develop the tool's clinician interface. The CHAMP tool is now ready for field testing.

The study objectives are to measure feasibility outcomes and efficacy of the tool in the identification of geriatric issues and development of care plan strategies.

Methods:

A total of 210 older adults (70+y) who have been referred to any kind of non-oncological surgery will be recruited from 4 centres -University Health Network, Sunnybrook Health Sciences Centre, St. Michael's Hospital and Mount Sinai Hospital. Older adults who agree to participate will be asked to provide information on sociodemographic characteristics and comfort with technology prior to completing the CHAMP tool. Subsequently, participants will be asked to complete the tool either prior to clinic (at home via internet) or in clinic (via iPad) prior to the participants' consultation with the clinician. Following completion of the CHAMP tool and prior to treatment decision making visit with the clinician, a member of the research team will provide the CHAMP results to the clinician. The clinician will be asked the proposed treatment plan and whether the patient is fit, vulnerable, or frail using standard definitions. Then, the clinician will be asked of whether the treatment plan intent is being modified based on the CHAMP tool. The CHAMP tool also contains evidence-based recommendations for clinicians on strategies to reduce risk and address geriatric domains. Surveys will be used to assess participants' and clinicians' satisfaction with the tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 years old and over who have been referred to any kind of non-oncological surgery
* Able to speak English
* Able to provide informed consent

Exclusion Criteria:

-

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Completeness of the CHAMP tool | Within one week from medical appointment
  Proportion of older adults who consented to the study who completed the CHAMP tool and had a discussion with the participants' physician about the CHAMP results.
Time to fill out the CHAMP tool | Within one week from medical appointment
  In minutes, recorded via user interaction logs which will include data such as user's actions and interactions with the actual interface such as clicks, point-an-select actions, use of back button, etc.), and whether the participant completed it alone or needed help.
Satisfaction with the CHAMP tool | Older adults - within one week of the participants' medical appointment. physicians - within one week of the last study patient.
  Measured via open-ended questions and a brief survey.

SECONDARY OUTCOMES:
Change in proposed treatment plan | Within 48 hours of the appointment with an older adults who has completed the CHAMP tool
  The impact of the CHAMP tool on proposed treatment plan will be measured through an adapted questionnaire which the investigators used in previous studies. It measures if treatment was changed at all (yes/no), and if changed, then modified intensity, alternate modality, best supportive care only, or other.
Changes in supportive care strategies | Within 48 hours of the appointment with an older adult who completed the CHAMP tool
  The impact of the the CHAMP tool on supportive care strategies will be measured through a survey that will be completed by the treating clinician. Additionally, the investigators will record the number of geriatric issues identified in the CHAMP summary and the number and type of recommendations provided to older adults and clinicians. The investigators will then review the charts of all older adults who completed CHAMP to abstract data on recommendations made by clinicians, referrals made to geriatrics and other health care providers, and other tests requested based on the recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Puts, PhD RN, Principal Investigator — University of Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the data available to other researchers